CLINICAL TRIAL: NCT06150742
Title: A Randomized, Placebo-controlled, Double-blind, Multi-center Study of the Safety and Efficacy of Niyad in Patients Undergoing Continuous Renal Replacement Therapy (CRRT) Who Cannot Tolerate Heparin or Are at a Higher Risk for Bleeding
Brief Title: Nafamostat Efficacy in Phase 3 Registrational CRRT Study
Acronym: NEPHRO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Talphera, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NYD301
Record Dates: First submitted 2023-11-21; First posted 2023-11-29 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2024-10

CONDITIONS: Acute Kidney Injury
Keywords: continuous renal replacement therapy; anticoagulation
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Niyad (Experimental): 1 mg/mL infusion of nafamostat mesylate
  Interventions: Device: Niyad (nafamostat mesylate)
- Placebo (Placebo Comparator): 0.9% saline infusion
  Interventions: Device: Placebo (0.9% NaCl)

INTERVENTIONS:
Device: Niyad (nafamostat mesylate) — Niyad (nafamostat mesylate) lyophilized
  Arms: Niyad
Device: Placebo (0.9% NaCl) — 0.9% NaCl
  Arms: Placebo

SUMMARY:
A prospective, randomized, placebo-controlled clinical study to investigate the safety and efficacy of Niyad (nafamostat mesylate) for anticoagulation of extracorporeal blood circulating through a dialysis filter in patients undergoing CRRT who cannot tolerate heparin or are at higher risk for bleeding.

DETAILED DESCRIPTION:
Patients in intensive care units with acute kidney injury are often too frail to undergo the rapid fluid shifts that accompany intermittent hemodialysis. Continuous renal replacement therapy (CRRT) allows a more gentle continual dialysis, more similar to regular kidney function. Anticoagulation of the CRRT circuit can reduce clotting of the filter, which can lead to less filter changes and possibly less transfusions. Niyad (nafamostat mesylate), an anticoagulant with an ultra-short half-life of 8 minutes, is approved for use in South Korea and Japan for anticoagulation of the CRRT circuit. For patients who cannot tolerate heparin or who are at a high risk of bleeding, nafamostat may be an optimal anticoagulant to infuse into the CRRT circuit as the short half-life should minimize patient exposure. The primary objective of this study is to measure the anticoagulation efficacy of Niyad in the CRRT circuit versus placebo. Evaluation of the safety of Niyad in patients undergoing CRRT versus placebo will also be performed.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring CRRT or undergoing CRRT initiated within the prior 48 hours
* Patients who cannot tolerate heparin or are at high risk of bleeding

Exclusion Criteria:

* Patients weighing less than 50 kg
* Patients receiving systemic anticoagulation
* Patients with active bleeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-08-15 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
mean post-filter activated clotting time (ACT) | 24 hours
  mean post-filter activated clotting time (ACT)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - University of California Los Angeles, Los Angeles, California
  - AdventHealth, Orlando, Florida
  - Henry Ford Health, Detroit, Michigan
  - University of New Mexico, Albuquerque, New Mexico
  - Northwell Health, Great Neck, New York
  - Mount Sinai, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Baylor University Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No